CLINICAL TRIAL: NCT04716595
Title: A Phase III Long Term Study of K-877 Extended Release Tablet-A Multicenter, Randomized, Open Label, Parallel Group Trial in Patients With Dyslipidemia With High TG-
Brief Title: A Phase III Long Term Study of K-877 Extended Release Tablet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-877-ER-03
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morning administration (Experimental): K-877 ER 0.2 mg/day morning administration (once daily)
  Interventions: Drug: K-877 ER 0.2 mg/day morning administration (once daily)
- evening administration (Experimental): K-877 ER 0.2 mg/day evening administration (once daily)
  Interventions: Drug: K-877 ER 0.2 mg/day evening administration (once daily)

INTERVENTIONS:
Drug: K-877 ER 0.2 mg/day morning administration (once daily) — K-877 ER 0.2 mg tablet
  Other Names: Pemafibrate ER 0.2 mg/day morning administration (once daily)
  Arms: morning administration
Drug: K-877 ER 0.2 mg/day evening administration (once daily) — K-877 ER 0.2 mg tablet
  Other Names: Pemafibrate ER 0.2 mg/day evening administration (once daily)
  Arms: evening administration

SUMMARY:
To investigate the safety and efficacy of K-877 Extended Release (ER) once daily for 52 weeks in the morning or evening in dyslipidema.The starting dose of the ER tablet will be 0.2 mg/day. If the efficacy is insufficient, it will investigate the safety and efficacy of 0.4 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia had to be age 20 years or older at written informed consent
2. Patients who have received dietary or exercise guidance from 12 weeks or more prior to Screening
3. Patients with the fasting serum TG >= 150 mg/dL twice consecutively at Screening

Exclusion Criteria:

1. Patients with a fasting serum TG > 1000 mg/dL at Screening
2. Patients who require administration of prohibited drugs during the clinical trial period after written informed consent
3. Patients with uncontrolled thyroid disease
4. Patients with type 1 diabetes and uncontrolled diabetes [HbA1c(NGSP) >= 10.0 % at Screening]
5. Patients with uncontrolled hypertension (SBP >= 160 mmHg or DBP >= 100 mmHg)
6. Patients with an AST or ALT three times the upper limit at Screening
7. Patients with an CK five times the upper limit at Screening
8. Patients with cirrhosis or those with biliary obstruction
9. Patients with acute myocardial infarction within 3 months before obtaining informed consent
10. Patients with heart failure class III or higher according to NYHA cardiac function classification
11. Patients with malignant tumor or those who are judged to have a high risk of recurrence
12. Patients with a history of serious drug allergies (anaphylactic shock, etc.)
13. Pregnant women, lactating women, women planning to become pregnant or lactating during the study period, or pregnant women who do not use specific contraceptive methods
14. Patients who have collected 400 mL or more of whole blood within 16 weeks, or 200 mL or more of whole blood within 4 weeks, or blood samples (plasma and platelet components) within 2 weeks before Screening
15. Patients who have received K-877 (pemafibrate)
16. Patients who participate in other clinical trials at the time of written informed consent and who received medication or who have received clinical trials other than placebo for less than 16 weeks
17. Patients who have been determined inappropriate by the investigator, etc

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Efficacy : Mean of percent change from baseline in fasting serum TG (mg/dL) at the time of final evaluation* and immediately before it * : Week 52 or at discontinuation | Final evaluation (Week 52 or at discontinuation) and immediately before it

SECONDARY OUTCOMES:
Efficacy : Mean of percent change from baseline in fasting serum Total Cholesterol (mg/dL) at the time of final evaluation* and immediately before it * : Week 52 or at discontinuation | Final evaluation (Week 52 or at discontinuation) and immediately before it
Efficacy : Mean of percent change from baseline in fasting serum LDL-C (mg/dL) at the time of final evaluation* and immediately before it * : Week 52 or at discontinuation | Final evaluation (Week 52 or at discontinuation) and immediately before it
Efficacy : Mean of percent change from baseline in fasting serum HDL-C (mg/dL) at the time of final evaluation* and immediately before it * : Week 52 or at discontinuation | Final evaluation (Week 52 or at discontinuation) and immediately before it
Efficacy : Mean of percent change from baseline in fasting serum non-HDL-C (mg/dL) at the time of final evaluation* and immediately before it * : Week 52 or at discontinuation | Final evaluation (Week 52 or at discontinuation) and immediately before it

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Saiseikai Futsukaichi Hospital, Fukuoka
  - National Hospital Organization Takasaki General Medical Center, Gunma
  - Hasegawa Medicine Clinic, Hokkaido
  - Japan Community Health care Organization Hokkaido Hospital, Hokkaido
  - Minami Akatsuka Clinic, Ibaraki
  - Saiseikai Yokohamashi Nanbu Hospital, Kanagawa
  - Kinugawa Cardiology Clinic, Osaka
  - Kyosokai AMC NISHI-UMEDA Clinic, Osaka
  - Medical corporation Tani clinic, Osaka
  - Shiraiwa medical clinic, Osaka
  - Cosmos medical corporation Aozora total clinic, Saitama
  - Akasaka Chuou Clinic, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Tokyo
  - Shimokitazawa Tomo Clinic, Tokyo

REFERENCES:
- [Result] Arai H, Yamashita S, Araki E, Yokote K, Tanigawa R, Saito A, Furukawa D, Suganami H, Ishibashi S. Long-Term Effects of Extended-Release Pemafibrate Tablets on Dyslipidemia and Safety in Triglyceridemic Patients: A Phase 3, Multicenter, Randomized, Open-Label, Parallel-Group Study. J Atheroscler Thromb. 2025 Aug 1;32(8):1006-1026. doi: 10.5551/jat.65350. Epub 2025 Feb 7. PMID 39924184